CLINICAL TRIAL: NCT04721015
Title: A Phase 1 First In Human Study Evaluating Safety And Efficacy Of ABBV-637 As Either Monotherapy Or In Combination In Adult Subjects With Relapsed And Refractory Solid Tumors
Brief Title: Study of Intravenous (IV) ABBV-637 Alone or in Combination With IV Docetaxel/Osimertinib to Assess Adverse Events and Change in Disease Activity in Adult Participants With Relapsed/Refractory (R/R) Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-111; 2020-004953-57 (EudraCT Number)
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors Cancer; Non Small Cell Lung Cancer (NSCLC)
Keywords: Advanced Solid Tumors Cancer; Non Small Cell Lung Cancer; NSCLC; Cancer; ABBV-637; Docetaxel; Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Docetaxel; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1: ABBV-637 Monotherapy (Experimental): Participants will receive escalating doses of ABBV-637 in 28-day cycles.
  Interventions: Drug: ABBV-637
- Part 2a: ABBV-637 + Docetaxel (Experimental): Participants will receive escalating doses of ABBV-637 in combination with docetaxel in 28-day cycles.
  Interventions: Drug: ABBV-637; Drug: Docetaxel
- Part 2b: ABBV-637 + Docetaxel (Experimental): Participants will receive ABBV-637 at dose determined in Part 2a in combination with docetaxel in 28-day cycles.
  Interventions: Drug: ABBV-637; Drug: Docetaxel
- Part 3a: ABBV-637 + Osimertinib (Experimental): Participants will receive escalating doses of ABBV-637 in combination with osimertinib in 28-day cycles.
  Interventions: Drug: ABBV-637; Drug: Osimertinib
- Part 3b: ABBV-637 + Osimertinib (Experimental): Participants will receive ABBV-637 at dose determined in Part 3a in combination with osimertinib in 28-day cycles.
  Interventions: Drug: ABBV-637; Drug: Osimertinib

INTERVENTIONS:
Drug: ABBV-637 — Intravenous (IV) Infusion
Drug: Docetaxel — Intravenous (IV) Infusion
  Arms: Part 2a: ABBV-637 + Docetaxel; Part 2b: ABBV-637 + Docetaxel
Drug: Osimertinib — Oral Tablets
  Arms: Part 3a: ABBV-637 + Osimertinib; Part 3b: ABBV-637 + Osimertinib

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. Non-Small Cell Lung Cancer (NSCLC) is a solid tumor, a disease in which cancer cells form in the tissues of the lung. The purpose of this study is to evaluate the safety and efficacy (how well the study drug works against the disease) of ABBV-637 alone or in combination with docetaxel/osimertinib in participants with solid tumors (NSCLC). Adverse events and change in disease activity will be assessed.

ABBV-637 is an investigational drug being developed for the treatment of solid tumors. Study consists of 3 parts - monotherapy dose escalation (Part 1), combination dose escalation and expansion (Parts 2a and 2b) with docetaxel and combination dose escalation and expansion (Parts 3a and 3b) with osimertinib. Approximately 109 adult participants with relapsed/refractory (R/R) solid tumors will be enrolled in approximately 30 sites across the world.

In Part 1, participants with solid tumors will receive intravenous (IV) ABBV-637 in 28-day cycles. In Part 2a and 2b, participants will receive IV ABBV-637 in combination with IV docetaxel in 28-day cycles. In Part 3a and 3b, participants will receive intravenous (IV) ABBV-637 in combination with daily oral tablets of osimertinib in 28-day cycle.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. Treatment effects will be monitored by medical assessments, blood tests, side effect reporting, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Histologic solid tumor diagnosis (Part 1).
* For Part 2 docetaxel combination therapy: EGFR WT expressing relapsed/refractory (R/R) non-small cell lung cancer (NSCLC) participants.
* For Part 3 osimertinib combination therapy: mutEGFR-expressing RR NSCLC participants.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* For Part 1 only - history of R/R disease that has progressed on all standard of care therapy.
* For Part 2 only - history of RR NSCLC that has progressed after treatment with platinum-based chemotherapy regimen and either immune checkpoint inhibitor or targeted therapy and may not have been treated with prior single agent chemotherapy.
* For Part 3 only - history of RR NSCLC that has progressed on osimertinib
* Meet the laboratory values as described in the protocol.

Exclusion Criteria:

* History (within 6 months) of congestive heart failure (defined as New York Heart Association, Class 2 or higher), ischemic cardiovascular event, cardiac arrhythmia requiring pharmacological or surgical intervention, pericardial effusion, or pericarditis.
* Unresolved Grade 2 or higher toxicities related to previous anticancer therapy except alopecia.
* For Part 3 only: History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, nor any evidence of active ILD or pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 3 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Percentage of Participants With Objective Response Rate (ORR) (Part 2 & 3) | Up to approximately 3 years
  ORR is defined as the percentage of participants with a confirmed response (CR) or partial response (PR) per investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response Rate (ORR) (Part 1) | Up to approximately 3 years
  ORR is defined as the percentage of participants with a confirmed response (CR) or partial response (PR) per investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of Response (DOR) for ABBV-637 Administered as Monotherapy (Part 1) | Up to approximately 12 months
  DOR is defined as the time from the initial response of CR/PR per investigator review according to RECIST version 1.1 criteria to the first occurrence of radiographic disease progression, clinical progression or death from any cause whichever occurs first.
Duration of Response (DOR) for ABBV-637 in Combination With Docetaxel and Osimertinib (Part 2 & 3) | Up to approximately 20 months
  DOR is defined as the time from the initial response of CR/PR per investigator review according to RECIST version 1.1 criteria to the first occurrence of radiographic disease progression, clinical progression or death from any cause whichever occurs first.
Progression-Free Survival (PFS) for ABBV-637 in Combination With Docetaxel and Osimertinib (Part 2 & 3) | Up to approximately 20 months
  PFS is defined as the time from the first dose of any study drug to a documented radiographic disease progression according to RECIST version 1.1 as determined by the investigator, clinical progression or death from any cause, whichever occurs earlier.
Overall Survival (OS) for ABBV-637 in Combination With Docetaxel and Osimertinib (Part 2 & 3) | Up to approximately 12 months after last dose of study drug
  OS is defined as the time from the first dose of any study drug until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (33):
- United States (6):
  - Dana-Farber Cancer Institute /ID# 231209, Boston, Massachusetts
  - Washington University-School of Medicine /ID# 225698, St Louis, Missouri
  - Carolina BioOncology Institute /ID# 225358, Huntersville, North Carolina
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 226145, Providence, Rhode Island
  - South Texas Accelerated Research Therapeutics /ID# 225359, San Antonio, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 225693, Fairfax, Virginia
- Australia (2):
  - Wollongong Hospital /ID# 228350, Wollongong, New South Wales
  - Austin Health /ID# 225638, Heidelberg, Victoria
- France (5):
  - AP-HM - Hopital de la Timone /ID# 225779, Marseille, Bouches-du-Rhone
  - Institut Bergonie /ID# 225778, Bordeaux, Gironde
  - Institut Curie /ID# 225829, Paris, Paris
  - Centre Georges François Leclerc /ID# 226760, Dijon
  - Institut Claudius Regaud /ID# 225780, Toulouse
- Israel (2):
  - Rambam Health Care Campus /ID# 225586, Haifa, H_efa
  - The Chaim Sheba Medical Center /ID# 225585, Ramat Gan, Tel Aviv
- Japan (5):
  - NHO Nagoya Medical Center /ID# 244412, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 225725, Kashiwa-shi, Chiba
  - Duplicate_National Hospital Organization Shikoku Cancer Center /ID# 240821, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center /ID# 240761, Fukuoka, Fukuoka
  - National Cancer Center Hospital /ID# 225724, Chuo-ku, Tokyo
- South Korea (4):
  - National Cancer Center /ID# 231887, Goyang-si, Gyeonggido
  - Asan Medical Center /ID# 231886, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 231888, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 233774, Seoul
- Spain (5):
  - Hospital Universitario Vall d'Hebron /ID# 225976, Barcelona, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 225975, Madrid, Madrid
  - Hospital Universitario 12 de Octubre /ID# 225977, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 226096, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 225978, Málaga, Malaga
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 243345, Kaohsiung City, Kaohsiung
  - National Cheng Kung University Hospital /ID# 225944, Tainan, Tainan
  - National Taiwan University Hospital - Hsinchu branch /ID# 243610, Hsinchu
  - Linkou Chang Gung Memorial Hospital /ID# 225946, Taoyuan

IPD SHARING:
Plan to Share IPD: No